CLINICAL TRIAL: NCT07262762
Title: A Post-marketing Real-world Study for Evaluating Effectiveness and Safety of Spartina® (Tirzepatide Manufactured by CinnaGen) in Patients With Obesity and Overweight
Brief Title: Spartina® (Tirzepatide) Effectiveness and Safety Evaluation
Status: Recruiting | Type: Observational
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Other Study IDs: TIR.CIN.AE.IV.04
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Obesity & Overweight
Keywords: obesity; overweight; tirzepatide
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to evaluate Effectiveness and safety of Spartina® (Tirzepatide) in male or female participants with obesity and overweight. The main questions which are aimed to be answered:

1. Is Spartina® (Tirzepatide) effective in the treatment of obesity and overweight?
2. Is Spartina® (Tirzepatide) safe in the treatment of obesity and overweight?

In this study, there is no comparison group. Participants receive Spartina® (Tirzepatide)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age
2. Willingness for signing and having signed the informed consent form
3. BMI ≥30 kg/m² or ≥27 kg/m² with ≥1 weight-related comorbidity

Exclusion Criteria:

1. Prior use of any GLP-1 agonist in the last 6 months
2. Type 1 diabetes mellitus
3. Any condition or circumstance that might pose a risk to the subject or interfere with the ability to acquire satisfactory clinical data
4. Pregnancy or breast-feeding
5. Personal or family history of medullary thyroid carcinoma (MTC) or patients with multiple endocrine neoplasia syndrome type 2 (MEN 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with ≥5% weight loss | day 0, 180

SECONDARY OUTCOMES:
Percent change in body weight from baseline | day 0, 90
Absolute change in body weight from baseline | day 0, 90
Percent change in body weight from baseline | day 0, 180
Absolute change in body weight from baseline | day 0, 180
Mean change in Body Mass Index from baseline | day 0, 90, 180
  24.9<BMI<30 and more than 30 are considered overweight and obesity, respectively. More BMI decrease is related to the better response.
Mean change in waist circumference from baseline | day 0, 90, 180
Proportion of patients with ≥5% weight loss | day 0, 90
Proportion of patients with ≥10% weight loss | day 0, 90, 180
Proportion of patients with ≥15% weight loss | day 0, 180
Assessment of the adverse events (including Treatment Emergent Adverse Events) | during study period
Assessment of immunogenicity at screening | day 0, 90, 180

CONTACTS AND LOCATIONS:
Locations (14):
- Iran (14):
  - Akbar Aliasgarzadeh Clinic, Tabriz, East Azerbaijan Province
  - Dr. Mohammadhossein Dabbaghmanesh Clinic, Shiraz, Fars
  - Behrang Motamed Clinic, Rasht, Gilan Province
  - Seyed Mojtaba Mehrdad Clinic, Rasht, Gilan Province
  - Mansoor Siavash Dastjerdi Clinic, Isfahan, Isfahan
  - Shokoofeh Bonakdaran Clininc, Mashhad, Khorasan Razavi
  - Sari Diabetes Research Center, Sari, Mazandaran
  - Alireza Esteghamati clinic, Tehran, Tehran Province
  - Farzad Hadaegh Clininc, Tehran, Tehran Province
  - Imam Khomeini Hospital, Tehran, Tehran Province
  - Iran University Endocrinology Research Center, Tehran, Tehran Province
  - Mohammadreza Mohajeri Tehrani Clininc, Tehran, Tehran Province
  - Khorshid Clinic, Yazd, Yazd Province
  - Hajieh Bibi Shahbazian Clinic, Ahvāz